CLINICAL TRIAL: NCT07164170
Title: An Open-label Phase II Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of ABSK043 in Combination With Glecirasib in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC) Harboring a KRAS G12C Mutation
Brief Title: A Phase 2 Clinical Study of Combination Therapy With ABSK043 and Glecirasib
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABSK043-201
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: ABSK043 in combination with Glecirasib (Experimental): This is an open-label phase 2 study with an escalation part and an expansion part.
  • Escalation Part: up to 50 previously treated patients with KRASG12C mutation. Does Escalation Cohort(Part A): up to 30previously treated patients with KRASG12C mutation.
  Dose Confirmation Cohort(Part B): up to 20previously treated patients with KRASG12C mutation.
  • Expansion Part: up to 36 treatment-naïve patients with KRASG12C mutation.
  Interventions: Drug: ABSK043 in combination with Glecirasib

INTERVENTIONS:
Drug: ABSK043 in combination with Glecirasib — Dose escalation cohort( Part A) ABSK043 150 mg BID in combination with Glecirasib 200 mg QD will be selected as the starting dose.
  Based on the accumulated safety data and PK profile, the Safety Review Committee (SRC), composed of the investigator and the sponsor, may discuss and agree to allow exploration of other possible doses.
  Dose confirmation cohort (Part B) and Expansion cohort Patients in dose confirmation cohort and expansion cohort will receive the recommended dose in dose escalation cohort and be evaluated for safety and preliminary anti-tumor activity.
  All patients will continue to receive combination therapy every 21 days until disease progression, death, loss to follow-up, withdrawal of consent, intolerable toxicity, investigator decision to discontinue treatment, or end of the study.

SUMMARY:
This is a multicenter, open-label phase 2 study that will enroll KRASG12C mutated patients with locally advanced or metastatic NSCLC, receiving treatment (ABSK043 in combination with Glecirasib) in a 21-day combination cycle.

DETAILED DESCRIPTION:
The study consists of an escalation part and an expansion part. The escalation part will evaluate the safety, tolerability, preliminary efficacy, and PK profile of different doses of ABSK043 in combination with Glecirasib, and the combination regimen recommended for the expansion part. The expansion part will further evaluate the safety, PK profile, and anti-tumor efficacy of ABSK043 in combination with Glecirasib at the one or more recommended dose (s).

Up to 86 patients with locally advanced or metastatic Non-small Cell Lung Cancer (NSCLC) are planned to be enrolled in the study.

* Escalation Part: up to 50 previously treated patients with KRASG12C mutation.
* Expansion Part: up to 36 treatment-naïve patients with KRASG12C mutation.

ELIGIBILITY:
Inclusion Criteria:

1. Prior to any protocol- specific procedures are performed, the patient should understand and voluntarily sign and date the written informed consent form.
2. Gender was not limited patients aged ≥18 years at the time of signing the informed consent.
3. Histologically or cytologically confirmed locally advanced, unresectable, or metastatic non-small cell lung cancer (NSCLC).

   For patients in the dose-escalation cohort (Part A) of the escalation part:

   Patients must have experienced disease progression following at least one line of prior standard systemic therapy, but no more than two lines of systemic therapy.

   For patients in the dose confirmation cohort (Part B) of the escalation part :
   1. Prior treatment requirements for patients in cohort (Part B) are the same as those for patients in (Part A);
   2. Documented or central laboratory test report confirmed that the tumor was PD-L1 expression positive (≥1%) .

   For patients in the expansion cohort of the expansion part :
   1. Patients who have not received prior systemic therapy for locally advanced or unresectable/metastatic disease;
   2. Central laboratory test report confirmed that the tumor was PD-L1 expression positive (≥1%) .
4. Tumor tissue or blood test report confirmed KRASG12C mutation.
5. Patients must have at least one measurable lesion as defined by RECIST v1.1.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0~1.
7. Expected survival time of ≥3 months.
8. Patients must have adequate organ and bone marrow function.

Exclusion Criteria:

1. Histological or cytological evidence of small cell lung cancer or neuroendocrine carcinoma components.
2. Toxicities from prior antitumor therapy have not returned to baseline or stabilized.
3. Patients with active brain metastases.
4. The patient currently has active interstitial lung disease.
5. Patients currently have active autoimmune disease or a history of autoimmune disease that may be at risk for recurrence.
6. Any condition requiring systemic treatment with corticosteroids.
7. Uncontrolled or significant cardiovascular disease.
8. Has a known human immunodeficiency virus (HIV) infection that is not well controlled.
9. Any evidence of severe or uncontrolled diseases or other factors which in the Investigator's opinion makes it undesirable for the patients to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-10-25 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of DLT | At the end of Cycle 1 (each cycle is 21 days)
  Dose-limiting toxicities
AEs | From the time the patient signs the informed consent form throughout the study and up to 90 days after the last dose of ABSK043 or 30 days after the last dose of Glecirasib, whichever occurs first, up to 30 months.
  Adverse events
SAEs | From the time the patient signs the informed consent form throughout the study and up to 90 days after the last dose of ABSK043 or 30 days after the last dose of Glecirasib, whichever occurs first, up to 30 months.
  Serious adverse events (SAEs)
AESIs AESIs | From the time the patient signs the informed consent form throughout the study and up to 90 days after the last dose of ABSK043 or 30 days after the last dose of Glecirasib, whichever occurs first, up to 30 months.
  Adverse events of special interest (AESIs)
ORR | From date of enrolment#Cycle1 Day1# until disease progression, death, loss to follow-up, withdrawal of consent, intolerable toxicity, investigator's decision to discontinue treatment, or end of study, whichever comes first, assessed up to 50 months.
  objective response rate

SECONDARY OUTCOMES:
Cmax | From the date of enrolment #Cycle1 Day1# to #Cycle7#, and for patients who discontinue treatment before cycle 7 (C7), PK sampling will be performed at the EOT visit and assessed up to 10 months
  Maximum observed concentration
AUC | From the date of enrolment #Cycle1 Day1# to #Cycle7#, and for patients who discontinue treatment before cycle 7 (C7), PK sampling will be performed at the EOT visit and assessed up to 10 months.
  area under the concentration-time curve
t1/2 t1/2 | From the date of enrolment #Cycle1 Day1# to #Cycle7#, and for patients who discontinue treatment before cycle 7 (C7), PK sampling will be performed at the EOT visit and assessed up to 10 months.
  elimination half-life
Vz/F | From the date of enrolment #Cycle1 Day1# to #Cycle7#, and for patients who discontinue treatment before cycle 7 (C7), PK sampling will be performed at the EOT visit and assessed up to 10 months.
  apparent volume of distribution
CL/F | From the date of enrolment #Cycle1 Day1# to #Cycle7#, and for patients who discontinue treatment before cycle 7 (C7), PK sampling will be performed at the EOT visit and assessed up to 10 months.
  apparent oral clearance
Cmax,ss | From the date of enrolment #Cycle1 Day1# to #Cycle7#, and for patients who discontinue treatment before cycle 7 (C7), PK sampling will be performed at the EOT visit and assessed up to 10 months.
  maximum observed concentration after multiple doses maximum observed concentration after multiple doses maximum observed concentration after multiple doses
Cmin,ss | From the date of enrolment #Cycle1 Day1# to #Cycle7#, and for patients who discontinue treatment before cycle 7 (C7), PK sampling will be performed at the EOT visit and assessed up to 10 months.
  minimum observed concentration after multiple doses
AUCtau,ss | From the date of enrolment #Cycle1 Day1# to #Cycle7#, and for patients who discontinue treatment before cycle 7 (C7), PK sampling will be performed at the EOT visit and assessed up to 10 months.
  area under the concentration-time curve after multiple doses
AR | From the date of enrolment #Cycle1 Day1# to #Cycle7#, and for patients who discontinue treatment before cycle 7 (C7), PK sampling will be performed at the EOT visit and assessed up to 10 months.
  accumulation ratio
tmax | From the date of enrolment #Cycle1 Day1# to #Cycle7#, and for patients who discontinue treatment before cycle 7 (C7), PK sampling will be performed at the EOT visit and assessed up to 10 months.
  time to maximum observed concentration
DOR DOR | From date of enrolment#Cycle1 Day1# until disease progression, death, loss to follow-up, withdrawal of consent, intolerable toxicity, investigator's decision to discontinue treatment, or end of study, whichever comes first, assessed up to 50 months.
  Duration of response
PFS | From date of enrolment#Cycle1 Day1# until disease progression, death, loss to follow-up, withdrawal of consent, intolerable toxicity, investigator's decision to discontinue treatment, or end of study, whichever comes first, assessed up to 50 months.
  Progression-free survival
DCR | From date of enrolment#Cycle1 Day1# until disease progression, death, loss to follow-up, withdrawal of consent, intolerable toxicity, investigator's decision to discontinue treatment, or end of study, whichever comes first, assessed up to 50 months.
  Disease control rate
TTP | From date of enrolment #Cycle1 Day1# until disease progression, assessed up to 50 months.
  Time to progression
OS | From date of enrolment#Cycle1 Day1# until disease progression, death, loss to follow-up, withdrawal of consent, intolerable toxicity, investigator's decision to discontinue treatment, or end of study, whichever comes first, assessed up to 50 months.
  Overall survival Overall survival Overall survival

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital & Guangxi Cancer Institude, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital Tongji Medical College of Hust, Wuhan, Hubei
  - Hunan Cancer Hospitial, Changsha, Hunan
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Central Hospital Affiliated to Shangdong First Medical University, Jinan, Shangdong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital Sichuan University, Chengdu, Sichuan